CLINICAL TRIAL: NCT04353440
Title: Association Between Sagittal Patellar Offset and Anterior Knee Pain After Multiradius Total Knee Replacement.
Brief Title: Association Between Sagittal Patellar Offset and Anterior Knee Pain in Total Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Orkhan Aliyev, Residents Doctor, Department of Orthopaedics and Traumatology, Principal investigator, M.D., Bezmialem Vakif University
Other Study IDs: 19590
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Primary Gonarthrosis, Bilateral; Knee Osteoarthritis; Knee Arthritis
Keywords: total knee arthroplasty; anterior knee pain; sagittal patellar offset
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study to evaluate whether the position of the sagittal patellar offset is a predictive factor for anterior knee pain in subjects having undergone bilateral multiradius total knee replacement.

DETAILED DESCRIPTION:
A prospective, observational study. A total of to 80 subjects requiring bilateral multiradius knee arthroplasty will be enrolled. Anterior femoral offset, femoral diameter and patellar offset will be measured by orthopaedic surgeons. In addition, Visual Analogue Scale Score, Oxford Knee Score, WOMAC, SF12 and SF36 will be evaluated postoperative in patients long-term follow up to see if there is a relationship between anterior femoral offset and anterior knee pain.In the direct lateral knee joint radiograph, the distance between the two parallel axis extending from both cortices of the femur is measured as "femoral diameter".The remaining length between the anterior axis and the maximum peak at the anterior of the prosthesis is considered as an "anterior femoral offset"[1]. Sagittal patellar offset defined by us as the ratio of the anterior femoral offset to the remaining distance between the maximum anterior point of the patella and the posterior vertex in the direct lateral knee joint radiography.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 50 years of age with primary severe gonarthrosis who will undergo total knee replacement

Exclusion Criteria:

* Patients with severe gonarthrosis, with a history of malignancy, with severe extraarticular deformity, with posttraumatic and septic arthritis sequel

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total knee arthroplasty due to severe gonarthrosis
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-04-23 (Estimated); Primary Completion 2025-04-23 (Estimated); Study Completion 2025-07-23 (Estimated)

PRIMARY OUTCOMES:
anterior patellar offset ratio | minimum 1 year
  The distance between the anterior cortex of the femur and the maximum peak at the anterior of the prosthesis is considered as an "anterior femoral offset"[1].Sagittal patellar offset defined by us as the ratio of the anterior femoral offset to the remaining distance between the maximum anterior point of the patella and the posterior vertex in the direct lateral knee joint radiography.

REFERENCES:
- [Background] Scott CEH, Clement ND, Yapp LZ, MacDonald DJ, Patton JT, Burnett R. Association Between Femoral Component Sagittal Positioning and Anterior Knee Pain in Total Knee Arthroplasty: A 10-Year Case-Control Follow-up Study of a Cruciate-Retaining Single-Radius Design. J Bone Joint Surg Am. 2019 Sep 4;101(17):1575-1585. doi: 10.2106/JBJS.18.01096. PMID 31483401